CLINICAL TRIAL: NCT04563923
Title: Treatment of Bullous Pemphigoid With Avdoralimab (IPH5401), an Anti-C5aR1 Monoclonal Antibody
Acronym: IPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-PP-13
Record Dates: First submitted 2020-09-17; First posted 2020-09-25 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — avdoralimab

STUDY DESIGN:
Intervention Model Description: It is a case-controlled, randomized, open-labelled, and multicenter phase II clinical trial. Four Dermatologic French centers (Nice, Marseille Nord, Marseille Timone and Montpellier university hospitals) specialized in the in the care of BP patients will be participating in the study. It is expected that forty subjects will be included in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (Experimental): Patients in this group will additionally receive 3 s.c. injections of avdoralimab every week during 12 weeks
  They receive 0.05% Clobetasol propionate cream as follows:
  * Patients of less than 45kg of body weight: 2 tubes of 10g/d
  * Patients of 45kg and above of body weight: 3 tubes of 10g/d Topical steroids will be applied every day until 15 days after the healing of the last bullous lesions
  Interventions: Drug: Avdoralimab (IPH5401)
- Conventional therapy (Other): Superpotent topical steroids are the gold standard treatment for BP. All patients will receive 0.05% Clobetasol propionate cream as follows:
  * Patients of less than 45kg of body weight: 2 tubes of 10g/d
  * Patients of 45kg and above of body weight: 3 tubes of 10g/d Topical steroids will be applied every day until 15 days after the healing of the last bullous lesions
  Interventions: Other: Control

INTERVENTIONS:
Drug: Avdoralimab (IPH5401) — Preparation of avdoralimab and preparation of the syringes are to be performed aseptically by site pharmacy qualified personnel.
  Arms: Drug
Other: Control — Superpotent topical steroids are the gold standard treatment for BP. All patients will receive 0.05% Clobetasol propionate cream as follows:
  * Patients of less than 45kg of body weight: 2 tubes of 10g/d
  * Patients of 45kg and above of body weight: 3 tubes of 10g/d Topical steroids will be applied every day until 15 days after the healing of the last bullous lesion
  Arms: Conventional therapy

SUMMARY:
The development of Auto Immune bullous Diseases (AIBD) results from a complex interaction between innate and adaptive immune systems. Bullous pemphigoid (BP), the most frequently encountered AIBD, predominantly affects elderly patients above 70 with an estimated incidence of 21.7 new cases/million/year in France.Interestingly, coversin, an anti-C5a and -leukotriene B4 small molecule, is currently used in a phase IIA clinical trial in BP patients (NCT04035733). However, although overall C5-blocking drugs are potentially interesting, they are likely to interfere with C5a-C5aR2-axis activation as well, a pathway that has recently proved protective in BP 12. The main objective is to investigate the clinical efficacy of an anti-C5aR1 antibody in addition to superpotent topical steroids compared to superpotent topical steroids alone in BP patients at 3 months.It is a case-controlled, randomized, open-labelled, and multicenter phase II clinical trial. Four Dermatologic French centers (Nice, Marseille Nord, Marseille Timone and Montpellier university hospitals) specialized in the in the care of BP patients will be participating in the study. It is expected that forty subjects will be included in this trial.

Conversely, a more targeted inhibition of C5a-C5aR1 axis might be more effective in BP, sparing the potentially protective effect of C5a-C5aR2 interaction.

Avdoralimab (IPH5401), a specific anti-C5aR1 monoclonal antibody, has already been credited of a good safety profile in the treatment of solid tumors and rheumatoid arthritis. The investigators hypothesize that avdoralimab might be a safe and effective treatment in BP patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ≥ 18 years of age at the time of signing the informed consent document
* Clinical diagnosis of BP confirmed by histology, immunohistochemistry and/or ELISA data
* Patient requiring a treatment by superpotent topical steroids
* Patients hospitalized for the treatment of their BP
* For female, only post-menopaused patients
* For male patients included in the study with partners of child bearing potential should agree to use highly effective contraception for the duration of the study and 6 months after the last dose of avdoralimab
* Signed informed consent document prior to any study related assessments/procedures being conducted
* Patient able to adhere to the study visit schedule and other protocol requirements
* Patient registered to the French Social Security

Exclusion Criteria:

* Patients requiring systemic steroids according to the physician in charge
* Contra indication to topical steroid
* Use of systemic steroids or any immunosuppressive drugs in the past 4 weeks
* Use of doxycycline or minocycline in the past 4 weeks
* Use of systemic rituximab or omalizumab or dupilimumab in the past 12 weeks
* Use of intravenous immunoglobulmins (IVIG) in the past 4 weeks
* Impossibility to come every week to receive the injection
* Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation
* Vulnerable people: pregnant or breast-feeding women, minors, adult under guardianship or deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Complete Clinical Remission | At 3 Months
  To investigate the clinical efficacy of an anti-C5aR1 antibody in addition to superpotent topical steroids compared to superpotent topical steroids alone in BP patients.The efficacy will be evaluated through the proportion of patients in complete clinical remission (CCR) at 3 months without any relapse during the study period. The CCR will be defined as the absence of new bullous and skin inflammatory lesions and absence of pruritus for at least 2 weeks.

SECONDARY OUTCOMES:
The delay | At 3 months
  To compare between the treatment groups the delay to complete clinical remission (CCR)
Initial Clinical Remission | At 3 months
  To compare between the treatment groups the delay to initial clinical remission (ICR)

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — CHU de Nice, Dermatologie
Locations (4):
- France (4):
  - CHU de Nice- Dermatologie, Nice, Alpes-Maritimes
  - APHM, Timone, Marseille, Bouche Du Rhône
  - APHM, Hôpital Nord, Marseille, Bouches Du Rhône
  - CHU Montpellier, Dermatologie, Montpellier, Herault

IPD SHARING:
Plan to Share IPD: Undecided